CLINICAL TRIAL: NCT00163943
Title: Neural Mechanisms Predisposing to Cardiovascular Risk in Individuals With the Metabolic Syndrome: Benefits of Dietary Weight Loss, Weight Loss Maintenance and Aerobic Exercise
Brief Title: Sympathetic Activity in Individuals With the Metabolic Syndrome: Benefits of Lifestyle Interventions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Bayside Health (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 7/05
Record Dates: First submitted 2005-09-12; First posted 2005-09-14 (Estimated); Last update posted 2007-08-01 (Estimated); Status verified 2005-09

CONDITIONS: Metabolic Syndrome X
Keywords: Metabolic syndrome; Sympathetic nervous system activity; Insulin sensitivity; weight loss; aerobic exercise
MeSH Terms: conditions — Metabolic Syndrome; Insulin Resistance; Weight Loss

INTERVENTIONS:
Behavioral: Dietary weight loss +/- aerobic exercise

SUMMARY:
An abdominal distribution of fat is associated with the greatest heart disease risk, because commonly, several risk factors of metabolic origin (high blood pressure, unfavourable cholesterol profile, elevated blood sugar, impaired insulin action) cluster in these individuals. When this occurs the condition is called the 'metabolic syndrome' (MetS). The cause of the MetS is yet to be fully elucidated. Increased activity of the nervous system resulting in enhanced release of the stress hormone 'norepinephrine', may be one mechanism by which adverse cardiovascular and metabolic sequelae of the MetS might be mediated. Dietary weight loss, and exercise are first-line treatments for the MetS and provide an opportunity to prevent or delay the development of type 2 diabetes and heart disease in this high risk group. However, there is a paucity of data regarding the effects of these lifestyle factors on the nervous system. Furthermore, it is also unknown whether active weight loss ('negative energy balance') or a stable lower weight (weight loss maintenance) is more important in modifying MetS components and nervous system activity. The aims of the proposed project are:

1. To determine whether dietary weight loss in combination with aerobic exercise is more beneficial than dietary weight loss alone in reducing nervous system activity and improving metabolic and cardiovascular parameters in middle-aged men and women with abdominal obesity and the MetS.
2. To determine whether weight loss maintenance four months after active weight loss is associated with a preservation of clinical benefits.
3. To study biological determinants of successful weight loss and weight loss maintenance.

DETAILED DESCRIPTION:
Background:

Autonomic dysfunction, namely increased sympathetic drive and reduced vagal tone, may participate in the pathogenesis and complications of the MetS. Weight loss and aerobic exercise are first-line therapeutic strategies that are known to be beneficial in lowering blood pressure, enhancing insulin action and preventing the development of type 2 diabetes. However, there is a paucity of data regarding their effects on sympathetic nervous system (SNS) activity. In a recently completed Pilot study in 22 MS subjects we demonstrated that moderate dietary weight loss (7% of initial body weight) is associated with marked reductions in whole-body norepinephrine spillover rate (by 43%, P= 0.005) and muscle sympathetic nervous activity (MSNA, by 15%, P=0.01). In the proposed project we wish to extend these observations by evaluating the clinical benefits of aerobic exercise and weight loss maintenance.

Aims:

1. To determine whether dietary weight loss in combination with aerobic exercise (WL + EX) is more beneficial than dietary weight loss alone (WL) in reducing SNS activity and improving cardiovascular and metabolic parameters in middle aged men and women with abdominal obesity and a diagnosis of the MetS.
2. To investigate the determinants of achieved weight loss, with a focus on the roles of SNS activity, b2-adrenoceptor polymorphisms, resting metabolic rate, plasma and interstitial adipocytokines.
3. To determine whether clinical benefits during active weight loss (negative energy balance) are sustained after a 4-month weight loss maintenance program and to investigate the determinants of successful weight loss maintenance (as above).
4. To examine the inter-relationships between SNS activity, insulin sensitivity, metabolic, anthropometric and haemodynamic parameters.

Subjects:

Sedentary men and women (n= 66) aged 45 to 65 years with a body mass index of 26 to 39 kg/m2, who fulfil Adult Treatment Panel III criteria for the MetS.

Study design:

Randomized, controlled, parallel design comparison of:

1. WL;
2. WL + EX; or
3. Control (no treatment).

Investigations will be performed at baseline, and at the end of 3-month lifestyle intervention, and a 4-month weight-maintenance program (WL and WL + EX groups).

Diets:

A modified version of the 'DASH' diet will be used at different caloric levels.

Exercise:

Bicycle riding, performed for 40 minutes on alternate days at a moderate intensity of 65% of maximum heart rate. Compliance will be assessed by VO2 max measurements.

Investigations:

SNS activity measurements (multiunit and single-unit microneurographic recordings of MSNA, whole-body norepinephrine spillover, and abdominal adipose tissue and skeletal muscle interstitial noradrenaline concentration determined by microdialysis) will be made before and during an oral glucose tolerance test, together with haemodynamic (calf blood flow measured by venous occlusion plethysmography) measurements. Changes in fat mass will be quantitated by DEXA scan. Metabolic measurements will include resting metabolic rate, insulin sensitivity, lipid profile, non-esterified fatty acids, plasma and interstitial adipokines/cytokines.

Clinical significance:

The proposed project will provide novel information about whole-body and regional sympathetic activity; the determinants of sympathetic activity and the relative clinical benefits of active weight loss, weight loss maintenance and aerobic exercise in middle-aged MetS subjects.

ELIGIBILITY:
Inclusion Criteria:

* Sixty six (33 male and 33 postmenopausal female) weight-stable (body mass index 26 to 39 kg/m2), sedentary, non-smoking subjects, aged 45 to 65 years will be recruited on the basis of having > 3 indices of the MetS as defined by Adult Treatment Panel (ATP) III criteria:

  * waist circumference > 102 cm for men and > 88 cm for women;
  * fasting plasma glucose level > 6.1 mmol/L, but nondiabetic (< 7.1 mmol/L);
  * fasting plasma triglyceride level > 1.69 mmol/L;
  * plasma high-density lipoprotein (HDL) level < 1.04 mmol/L (males) and < 1.29 mmol/L (females);
  * supine resting blood pressure > 130/85 mmHg and < 165/105 mmHg, at least 4 weeks off blood pressure lowering medications.

Exclusion Criteria:

Exclusion criteria will comprise:

* A history of diabetes, secondary hypertension, sleep apnoea, cardiovascular, cerebrovascular, renal, liver, or thyroid disease
* Inability to cease medications which may affect measured parameters
* Inability or contraindication to exercise

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2005-04; Study Completion 2007-12 (Estimated)

PRIMARY OUTCOMES:
Whole-body sympathetic activity
Muscle sympathetic activity

SECONDARY OUTCOMES:
Insulin sensitivity
Lipid profile
Adipocytokines
Blood pressure
Baroreflex function
Forearm and calf blood flow

CONTACTS AND LOCATIONS:
Overall Officials: Nora E Straznicky, BPharm, PhD, MPH, Principal Investigator — Baker Heart Research Institute
Locations (1):
- Baker Heart Research Institute, Melbourne, Victoria, Australia

REFERENCES:
- [Derived] Khan AA, Mundra PA, Straznicky NE, Nestel PJ, Wong G, Tan R, Huynh K, Ng TW, Mellett NA, Weir JM, Barlow CK, Alshehry ZH, Lambert GW, Kingwell BA, Meikle PJ. Weight Loss and Exercise Alter the High-Density Lipoprotein Lipidome and Improve High-Density Lipoprotein Functionality in Metabolic Syndrome. Arterioscler Thromb Vasc Biol. 2018 Feb;38(2):438-447. doi: 10.1161/ATVBAHA.117.310212. Epub 2017 Dec 28. PMID 29284607
- [Derived] Nestel PJ, Straznicky N, Mellett NA, Wong G, De Souza DP, Tull DL, Barlow CK, Grima MT, Meikle PJ. Specific plasma lipid classes and phospholipid fatty acids indicative of dairy food consumption associate with insulin sensitivity. Am J Clin Nutr. 2014 Jan;99(1):46-53. doi: 10.3945/ajcn.113.071712. Epub 2013 Oct 23. PMID 24153346